CLINICAL TRIAL: NCT01040598
Title: Identifying Responders to Xolair (Omalizumab) Using Eosinophilic Esophagitis as a Disease Model
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: O & O Alpan LLC (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EE001
Record Dates: First submitted 2009-12-27; First posted 2009-12-29 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic Esophagitis; Xolair; Omalizumab; Esophagitis; Eosinophils; monoclonal antibody
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophagitis | interventions — Omalizumab

INTERVENTIONS:
Biological: Omalizumab — Omalizumab, an anti-IgE monoclonal antibody is dosed on the basis of subject's weight and IgE levels. It is administered as a subcutaneous injection every 2 weeks or 4 weeks based on the total dose required.
  Other Names: Xolair

SUMMARY:
Eosinophilic Esophagitis(EoE) is a condition characterized commonly by vomiting, nausea, epigastric pain, dysphagia, heartburn and food impaction among other gastrointestinal symptoms along with obstructive esophageal symptoms in both pediatric and adult population. The pathology of this disease is postulated to be allergy mediated and the incidence of this disease is seen to parallel an increase in the incidence of allergies and asthma.

Most of the current therapies for EoE are directed at decreasing esophageal allergic inflammation and mirror the treatment options for allergic asthma. Swallowed corticosteroids and elimination diets or elemental diets have shown variable efficacy is improving symptoms. However, specific pathophysiologic mechanism of EoE is still largely unknown and there is no definitive treatment that completely resolves symptoms and histological findings. Omalizumab is a recently developed anti-IgE antibody that has been shown to decrease the use of inhaled and oral corticosteroids and improve asthma related symptoms in patients with allergic asthma. In this study, Eosinophilic esophagitis is being used as a disease model to study the mechanism of action of monoclonal Anti-IgE antibody in vivo. The resolution of symptoms clinically, and histological changes (and improvements) in response to treatment with Xolair (omalizumab) in patients suffering from EoE will be determined. The primary objective of this open label, study is to determine mucosal markers that will predict responders to Omalizumab (Xolair).

DETAILED DESCRIPTION:
This is an open label mechanistic study to learn about the effect of Omalizumab on the clinical symptoms and immunohistological findings in established cases of EoE. The dosage for Omalizumab will be based on patient's body weight and baseline IgE level. Omalizumab will be administered subcutaneously every 2 or 4 weeks for total duration of 12 weeks. At enrollment, subjects will have EGD with biopsies performed to confirm diagnosis of EoE and further histologic analysis and special staining. Blood will be drawn for baseline testing and monthly for safety labs. At the end of the 12 week period, repeat endoscopy will be performed and biopsies taken to stain again for various mucosal markers like IgE, IL-13, IL-5 and Tryptase. The patients will be followed for response to therapy with regards to resolution of symptoms and improvement in histology findings on biopsy.

ELIGIBILITY:
Inclusion criteria

* Established diagnosis of eosinophilic esophagitis, determined by eosinophils >15/high power field in the distal esophagus and/or microabscesses.
* Patients should be on therapy either by food avoidance or swallowed steroids, with no change in the food avoidance and steroid dose during therapy.
* One active symptom of disease (epigastric pain, vomiting, nausea, dysphagia or heartburn) at least 2 days of the week.
* Failed response to proton pump inhibitors or a negative ph probe test or Negative impedance study.
* Males and females between ages 12-76 years.

Exclusion criteria

* Patients with gastrointestinal reflux disease.
* Eosinophilic disease in the stomach or duodenum.
* Peripheral eosinophil counts >1500 (hyper eosinophilic syndrome).
* Women of childbearing potential not using two forms of contraception method(s) including but not limited to condoms, diaphragm, oral contraceptive pills, other hormonal methods, intrauterine device or tubal ligation and vasectomy, as well as women who are breastfeeding
* Known sensitivity to study drug(s) or class of study drug(s).
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study (specify as required).
* Use of any other investigational agent in the last 30 days.
* Use of systemic or inhaled steroids within the past 1 month.
* History of malignancy.
* Require chronic immunosuppressive therapy including cyclosporine, methotrexate, etc.
* Have been treated with Xolair within the 12 months prior to screening.
* Patients with eosinophilic esophagitis in remission on swallowed steroids.
* Patients with asthma taking inhaled steroids.
* Serum IgE levels < 30 IU/l or > 700 IU/l

Ages: 12 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-06; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Our primary objective is to determine markers that will predict responders to Omalizumab(Xolair) | 12 weeks

SECONDARY OUTCOMES:
Secondary objectives will be determining the immunological changes in the tissue before and after treatment with Xolair (omalizumab) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oral Alpan, MD, Principal Investigator — O & O Alpan LLC
Locations (1):
- O & O Alpan LLC, Springfield, Virginia, United States

REFERENCES:
- [Derived] Loizou D, Enav B, Komlodi-Pasztor E, Hider P, Kim-Chang J, Noonan L, Taber T, Kaushal S, Limgala R, Brown M, Gupta R, Balba N, Goker-Alpan O, Khojah A, Alpan O. A pilot study of omalizumab in eosinophilic esophagitis. PLoS One. 2015 Mar 19;10(3):e0113483. doi: 10.1371/journal.pone.0113483. eCollection 2015. PMID 25789989